CLINICAL TRIAL: NCT02659020
Title: A Phase 1b (Open-Label)/Phase 2 (Randomized, Double-Blinded) Study Evaluating Gemcitabine and Docetaxel With or Without Olaratumab in the Treatment of Advanced Soft Tissue Sarcoma
Brief Title: A Study of Olaratumab (LY3012207) in Participants With Advanced Soft Tissue Sarcoma
Acronym: ANNOUNCE 2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15839; I5B-MC-JGDL (Other: Eli Lilly and Company); 2015-001316-34 (EudraCT Number)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Gemcitabine; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel (Experimental): Participants received intravenous infusions of olaratumab 15 milligrams per kilogram (mg/kg) on days 1, 8 plus gemcitabine 900 milligrams per meter square (mg/m^2) on days 1, 8 plus docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
  Interventions: Drug: Olaratumab; Drug: Gemcitabine; Drug: Docetaxel
- Phase 1b: Cohort 2 overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel (Experimental): Participants received intravenous infusions of olaratumab 20 mg/kg on days 1, 8 in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met (cohort 2). Following a protocol amendment, additional participants were enrolled into this group to confirm the safety of the 20 mg/kg dose level prior to opening the Phase 2 (cohort 2 expansion).
  Interventions: Drug: Olaratumab; Drug: Gemcitabine; Drug: Docetaxel
- Phase 2: Olaratumab + Gemcitabine + Docetaxel (Experimental): Participants received intravenous infusions of olaratumab loading dose 20 mg/kg on days 1, 8 of cycle 1 followed by 15 mg/kg on days 1, 8 of all subsequent cycles in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met. This cohort is a combination of participants who never received olaratumab (olaratumab-naive) and who received commercially available olaratumab (olaratumab pre-treated) prior to enrollment.
  Interventions: Drug: Olaratumab; Drug: Gemcitabine; Drug: Docetaxel
- Phase 2: Placebo + Gemcitabine + Docetaxel (Placebo Comparator): Participants received intravenous infusions of placebo on days 1, 8 in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met. This cohort is a combination of participants who never received olaratumab (olaratumab-naive) and who received commercially available olaratumab (olaratumab pre-treated) prior to enrollment.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207; IMC-3G3
  Arms: Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel; Phase 1b: Cohort 2 overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel; Phase 2: Olaratumab + Gemcitabine + Docetaxel
Drug: Gemcitabine — Administered IV
  Other Names: LY188011; Gemzar
Drug: Docetaxel — Administered IV
Drug: Placebo — Administered IV
  Arms: Phase 2: Placebo + Gemcitabine + Docetaxel

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of two anti-cancer drugs (gemcitabine and docetaxel) with and without the study drug known as olaratumab in participants with advanced soft tissue sarcoma (STS) or STS that has spread to another part(s) of the body.

ELIGIBILITY:
Inclusion Criteria:

* The participant may have no more than 2 prior lines of systemic therapies (neoadjuvant and adjuvant therapies will not be considered as a prior line of therapy) for advanced or metastatic disease and is suitable to receive gemcitabine and docetaxel therapy. All previous therapies must have completed ≥ 3 weeks (21 days) prior to first dose of study drug.
* In the Phase 2 part, prior olaratumab/doxorubicin combination therapy in 1 prior treatment line is allowed.

  * Prior olaratumab therapy must have been received with doxorubicin as indicated on the olaratumab label.
  * Prior olaratumab therapy must have included at least 2 full cycles of olaratumab/doxorubicin (that is, a minimum of 4 doses of olaratumab).
  * Participants, who completed at least 2 cycles of combination olaratumab/doxorubicin therapy then discontinued doxorubicin due to toxicity or maximum dosing and proceeded to olaratumab monotherapy, are eligible.
  * The most recent dose of olaratumab must have been received within 180 days of randomization in this study.
* Availability of tumor tissue is mandatory for study eligibility. The participant must have consented to provide archived formalin-fixed paraffin-embedded tumor tissue or be subject to a pre-treatment re-biopsy of primary or metastatic tumor tissue for future central pathology review and translational research (if archived tissue is unavailable).
* The participant has adequate hematologic, organ, and coagulation function within 2 weeks (14 days) prior to enrollment (Phase 1b) or randomization (Phase 2).

Exclusion Criteria:

* The participant is diagnosed with gastrointestinal stromal tumor (GIST) or Kaposi sarcoma.
* The participant has active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of enrollment (Phase 1b) or randomization (Phase 2). Participants with a history of a CNS metastasis previously treated with curative intent (for example, stereotactic radiation or surgery) that have not progressed on follow-up imaging, have been asymptomatic for at least 60 days, and are not receiving systemic corticosteroids and or/anticonvulsants, are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before enrollment (Phase 1b) /randomization (Phase 2) to rule out brain metastasis.
* The participant has received prior treatment with gemcitabine or docetaxel. Note: Participants previously enrolled in the I5B-MC-JGDJ (NCT02451943) or any other blinded study with olaratumab are not eligible to participate in this trial.
* The participant has electively planned or will require major surgery during the course of the study.
* Females who are pregnant or breastfeeding.
* The participant has an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (48):
- United States (21):
  - UCLA Medical Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Georgia Cancer Specialists PC, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University Medical School, St Louis, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Monter Cancer Center, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma Cancer Specialists & Research Institute, LLC, Tulsa, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Helios Klinikum Bad Saarow, Bad Saarow, Brandenburg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - HELIOS Klinikum Berlin-Buch, Berlin
- Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz, Szolnok, Hungary
- Israel (4):
  - Sheba Medical Center, Tel Litwinsky, Ramat Gan
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Fondazione Piemonte l'Oncologia-Istituto Ricerca Cura Cancro, Candiolo, Torino
  - Humanitas Gradenigo, Torino
- Centrum Onkologii-Instytut im Marii Sklodowskiej-Curie, Warsaw, Poland
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (4):
  - University College Hospital - London, London, Greater London
  - Royal Marsden NHS Trust, London, Greater London
  - Clatterbridge Cancer Centre, Bebbington, Merseyside
  - Western General Hospital, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Olaratumab (LY3012207) in Participants With Advanced Soft Tissue Sarcoma (ANNOUNCE-2) — https://trials.lillytrialguide.com/en-US/trial/3Jz0lQ8yUE2Q42EWCOQKWq

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause.
Groups:
- Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel: Participants received intravenous infusions of olaratumab 20 mg/kg on days 1, 8 in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
- Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel: Following a protocol amendment, additional participants were enrolled into this group to confirm the safety of the 20 mg/kg dose level prior to opening the Phase 2. Participants received intravenous infusions of olaratumab 20 milligrams per kilogram (mg/kg) on days 1, 8 plus gemcitabine 900 milligrams per meter square (mg/m^2) on days 1, 8 plus docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
- Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive): This cohort included participants who never received olaratumab prior to enrollment. Participants received intravenous infusions of olaratumab loading dose 20 mg/kg on days 1, 8 of cycle 1 followed by 15 mg/kg on days 1, 8 of all subsequent cycles in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
- Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated): This cohort included participants who received commercially available olaratumab prior to enrollment. Participants received intravenous infusions of olaratumab loading dose 20 mg/kg on days 1, 8 of cycle 1 followed by 15 mg/kg on days 1, 8 of all subsequent cycles in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
- Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive): This cohort included participants who never received olaratumab prior to enrollment. Participants received intravenous infusions of placebo on days 1, 8 in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
- Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated): This cohort included participants who received commercially available olaratumab prior to enrollment. Participants received intravenous infusions of placebo on days 1, 8 in combination with gemcitabine 900 mg/m^2 on days 1, 8 and docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Started | 21 | 18 | 15 | 81 | 46 | 86 | 43
Received at Least 1 Dose of Study Drug | 21 | 18 | 15 | 81 | 45 | 86 | 43
Completed | 18 | 15 | 14 | 65 | 40 | 75 | 35
Not Completed | 3 | 3 | 1 | 16 | 6 | 11 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1 | 6 | 1 | 5 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 3 | 3 | 6 | 3
Not completed — Progressive Disease | 0 | 0 | 0 | 4 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants from phase 1b/2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Total
Number analyzed (Participants) | 21 | 18 | 15 | 81 | 46 | 86 | 43 | 310
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 20 | 12 | 6 | 66 | 27 | 66 | 30 | 227
  >=65 years | 1 | 6 | 9 | 15 | 19 | 20 | 13 | 83
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 7 | 48 | 28 | 58 | 28 | 188
  Male | 10 | 10 | 8 | 33 | 18 | 28 | 15 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 1 | 8 | 4 | 6 | 4 | 28
  Not Hispanic or Latino | 16 | 18 | 11 | 71 | 39 | 73 | 36 | 264
  Unknown or Not Reported | 0 | 0 | 3 | 2 | 3 | 7 | 3 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 3 | 2 | 2 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 2 | 0 | 1 | 8 | 1 | 2 | 14
  White | 15 | 10 | 13 | 61 | 30 | 70 | 34 | 233
  More than one race | 6 | 5 | 0 | 15 | 3 | 10 | 3 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 11
  United States | 10 | 14 | 14 | 29 | 36 | 28 | 30 | 161
  Poland | 0 | 0 | 0 | 6 | 0 | 2 | 0 | 8
  United Kingdom | 0 | 0 | 0 | 11 | 3 | 12 | 5 | 31
  Italy | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 6
  Israel | 0 | 0 | 0 | 4 | 3 | 7 | 4 | 18
  France | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 5
  Australia | 0 | 0 | 1 | 6 | 0 | 2 | 0 | 9
  Germany | 0 | 0 | 0 | 7 | 4 | 11 | 2 | 24
  Spain | 11 | 4 | 0 | 9 | 0 | 11 | 2 | 37

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicity (DLT)
Description: A Dose Limiting Toxicity is defined as an Adverse Event (AE) that is likely related to the study medication or combination, and fulfils any one of the following criteria, graded according to the NCI-CTCAE Version 4.0:
  1. Febrile neutropenia with documented Grade ≥3 infection or sepsis
  2. Grade 4 neutropenia lasting 7 days or longer.
  3. Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia complicated by hemorrhage.
  4. Nonhematologic Grade ≥3 toxicity, except for toxicities such as nausea, vomiting, transient electrolyte abnormalities, or diarrhoea that can be controlled with optimal medical management within 48 hours.
Time Frame: Cycle 1 (Up To 21 Days)
Population: Phase 1b: All participants who received at least one dose of Olaratumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 21 | 18 | 15
Participants | 1 | 4 | 3

2. Primary Outcome: Phase 2: Overall Survival (OS) (Olaratumab-Naive)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. For each participant who is not known to have died as of the data-inclusion cut-off date for a particular analysis, overall survival duration was censored for that analysis at the date of last prior contact.
Time Frame: Baseline to Date of Death Due to Any Cause (Up To 38 Months)
Population: Phase 2: All randomized participants (including the censored participants). Number of participants censored in "Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) =30," "Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) =28."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive)
Number analyzed (Participants) | 81 | 86
Months | 16.76 [15.28 to 25.40] | 18.04 [13.17 to 22.90]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Test type: Superiority; p = 0.775, Log Rank — Stratified by number of prior systemic therapies for locally advanced or metastatic disease (0 vs ≥1), histological tumor type (leiomyosarcoma vs non-leiomyosarcoma), and Eastern Cooperative Oncology Group Performance Status (ECOG PS) (0 vs1); Hazard Ratio (HR) = 0.945, 95% CI 2-sided [0.639 to 1.397] — Stratified by number of prior systemic therapies for locally advanced or metastatic disease (0 vs ≥1), histological tumor type (leiomyosarcoma vs non-leiomyosarcoma), and ECOG PS (0 vs1)

3. Secondary Outcome: Phase 1b: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Olaratumab
Description: Cmax of Olaratumab.
Time Frame: Pre-dose, 5 minutes (min), 1, 4, 4.5, 24, 96, 168, 336 hours (h) post-dose on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 3 Day 1, Cycle 3 Day 8
Population: Phase 1b: All participants who received at least one dose of Olaratumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 20 | 33
micrograms per milliliter (μg/mL)
  Cycle 1 (Day 1): number analyzed (Participants) | 19 | 33
  Cycle 1 (Day 1) | 432 (24) | 572 (25)
  Cycle 1 (Day 8) | 460 (25) | 697 (20)
  Cycle 3 (Day 1): number analyzed (Participants) | 14 | 23
  Cycle 3 (Day 1) | 523 (38) | 644 (20)
  Cycle 3 (Day 8): number analyzed (Participants) | 14 | 22
  Cycle 3 (Day 8) | 513 (21) | 689 (20)

4. Secondary Outcome: Phase 1b: PK: Minimum Serum Concentration (Cmin) of Olaratumab
Description: Cmin of Olaratumab.
Time Frame: Pre-dose, 5 min, 1, 4, 4.5, 24, 96, 168, 336 h post-dose on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 3 Day 1
Population: Phase 1b: All participants who received at least one dose of Olaratumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 20 | 31
μg/mL
  Cycle 1 (Day 1) | 95.9 (37) | 142 (38)
  Cycle 1 (Day 8): number analyzed (Participants) | 19 | 30
  Cycle 1 (Day 8) | 64.3 (64) | 93.3 (47)
  Cycle 3 (Day 1): number analyzed (Participants) | 14 | 22
  Cycle 3 (Day 1) | 137 (40) | 252 (36)

5. Secondary Outcome: Phase 1b: PK: Elimination Half-Life (T1/2) of Olaratumab
Description: T1/2 of Olaratumab.
Time Frame: Pre-dose, 5 min, 1, 4, 4.5, 24, 96, 168, 336 h post-dose on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 3 Day 1, Cycle 3 Day 8
Population: Phase 1b: All participants who received at least one dose of Olaratumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 19 | 33
days
  Cycle 1 (Day 1) | 4.60 (34) | 4.29 (28)
  Cycle 1 (Day 8) | 6.25 (25) | 6.62 (27)
  Cycle 3 (Day 1): number analyzed (Participants) | 14 | 23
  Cycle 3 (Day 1) | 5.17 (36) | 6.36 (41)
  Cycle 3 (Day 8): number analyzed (Participants) | 14 | 21
  Cycle 3 (Day 8) | 5.82 (30) | 6.39 (32)

6. Secondary Outcome: Phase 1b/2: PK: Cmax of Gemcitabine
Description: Cmax of Gemcitabine.
Time Frame: Day 8 of Cycle 1 (end of infusion, 1, 2, 4, 24 hours post-infusion)
Population: Phase 1b/2: All participants who received at least one dose of Gemcitabine and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel | Phase 2: Placebo + Gemcitabine + Docetaxel
Number analyzed (Participants) | 18 | 24 | 87 | 88
μg/mL | 2.79 (70) | 3.49 (50) | 3.01 (122) | 2.35 (105)

7. Secondary Outcome: Phase 1b/2: PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC[0-∞]) of Gemcitabine
Description: AUC[0-∞] of Gemcitabine
Time Frame: Day 8 of Cycle 1 (end of infusion, 1, 2, 4, 24 hours post-infusion)
Population: Phase 1b/2: Zero participants analysed. Due to short half-life of Gemcitabine, there was insufficient quantifiable data in the elimination phase to calculate AUC[0-∞] for any of the participants.
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel | Phase 2: Placebo + Gemcitabine + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Phase 1b/2: PK: Cmax of Docetaxel
Description: Cmax of Docetaxel.
Time Frame: 5 min, 1, 3, 24, 48 h post-dose on Cycle 1 Day 8
Population: Phase 1b/2: All participants who received at least one dose of Docetaxel and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel | Phase 2: Placebo + Gemcitabine + Docetaxel
Number analyzed (Participants) | 18 | 30 | 71 | 73
Nanograms per milliliter | 903 (143) | 1110 (84) | 1030 (134) | 827 (102)

9. Secondary Outcome: Phase 1b/2: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC [0-∞]) of Docetaxel
Description: AUC [0-∞] of Docetaxel.
Time Frame: 5 min, 1, 3, 24, 48 h post-dose on Cycle 1 Day 8
Population: Phase 1b/2: All participants who received at least one dose of Docetaxel and had evaluable PK data. For phase 2, zero participants analysed due to data not collected for AUC [0-∞] of Docetaxel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Overall - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel | Phase 2: Placebo + Gemcitabine + Docetaxel
Number analyzed (Participants) | 7 | 18 | 0 | 0
nanograms*hours per milliliter | 4440 (103) | 2990 (83) |  |

10. Secondary Outcome: Phase 1b/2: Population PK: Clearance of Olaratumab
Description: Population PK: Clearance of Olaratumab
Time Frame: Cycle 1-19: Pre-dose, 5 min, 1, 4, 4.5, 24, 96, 168, 336 h post-dose on days 1, 8
Population: Phase 1b/2: All participants who received at least one dose of Olaratumab and had evaluable PK data. Phase 1b and phase 2 participants olaratumab PK data was planned to be pooled for the population PK analysis and compared to a validated PK model to confirm that PK parameters were similar to analyses from previous olaratumab studies.
Measure: Mean (95% Confidence Interval); unit: Liter Per Hour
Groups:
- Olaratumab + Gemcitabine + Docetaxel: Participants received intravenous infusions of olaratumab on days 1, 8 (phase 1: 15 or 20 mg/kg; phase 2: 20 mg/kg only in cycle 1 and 15 mg/kg in subsequent cycles) plus gemcitabine 900 mg/m^2 on days 1, 8 plus docetaxel 75 mg/m^2 on day 8 of a 21-day cycle until disease progression, unacceptable toxicity, death, or other discontinuation criteria were met.
Arm/Group | Olaratumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 178
Liter Per Hour | 0.0186 [0.0175 to 0.0192]

11. Secondary Outcome: Phase 1b/2: Population PK: Volume of Distribution at Steady State (Vss) of Olaratumab
Description: The Vss is the sum of central volume of distribution (V1) + peripheral volume of distribution (V2).
Time Frame: Cycle 1-19: Pre-dose, 5 min, 1, 4, 4.5, 24, 96, 168, 336 h post-dose on days 1, 8
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Olaratumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 178
Liter | 5.14 [4.68 to 5.54]

12. Secondary Outcome: Phase 2: Overall Survival (Olaratumab Pre-Treated)
Description: as for outcome 2
Time Frame: Baseline to Date of Death Due to Any Cause (Up To 38 Months)
Population: Phase 2: All randomized participants (including the censored participants). Number of participants censored in "Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-Treated) = 20," "Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-Treated) =15."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 46 | 43
Months | 19.84 [14.19 to NA] — There were not enough events to estimate the upper confidence limit. | 17.31 [10.81 to 20.30]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Test type: Superiority; p = 0.148, Log Rank — Stratified by number of prior systemic therapies for locally advanced or metastatic disease (0 vs ≥1), histological tumor type (leiomyosarcoma vs non-leiomyosarcoma), and ECOG PS (0 vs1); Hazard Ratio (HR) = 0.667, 95% CI 2-sided [0.385 to 1.158] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first date of radiologic disease progression (as defined by Response Evaluation Criteria In Solid Tumors, Version 1.1 [RECIST v.1.1]) or death due to any cause. Progressive disease (PD) was defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Participants who have neither progressed nor died were censored at the day of their last radiographic tumor assessment, if available, or date of randomization if no post-baseline radiographic assessment is available.
Time Frame: Baseline to Objective Disease Progression or Death from Any Cause (Up To 38 Months)
Population: Phase 2: All randomized participants (including the censored participants). Number of participants censored in "Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive)=20" "Placebo + Gemcitabine + Docetaxel (Olaratumab-naive)=21," "Olaratumab + Gemcitabine + Docetaxel (Olaratumab pre-treated)=12," "Placebo + Gemcitabine + Docetaxel (Olaratumab pre-treated)=16."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 81 | 86 | 46 | 43
Months | 7.62 [5.13 to 8.54] | 4.37 [2.86 to 6.87] | 5.45 [2.76 to 8.71] | 4.17 [2.20 to 6.90]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Test type: Superiority; p = 0.055, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.692, 95% CI 2-sided [0.476 to 1.007] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Test type: Superiority; p = 0.482, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.828, 95% CI 2-sided [0.490 to 1.398]

14. Secondary Outcome: Phase 2: Percentage of Participants With a Complete or Partial Response (Objective Response Rate [ORR])
Description: ORR is the best overall tumor response of complete response (CR) or partial response (PR) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Baseline to Objective Disease Progression or Start of New Anti-Cancer Therapy (Up To 38 Months)
Population: Phase 2: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 81 | 86 | 46 | 43
Percentage of participants | 32.1 [22.2 to 43.4] | 23.3 [14.8 to 33.6] | 30.4 [17.7 to 45.8] | 14 [5.3 to 27.9]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Test type: Superiority; p = 0.1891, Exact Mantel-Haenszel test — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 1.589, 95% CI 2-sided [0.794 to 3.179] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Test type: Superiority; p = 0.0642, Exact Mantel-Haenszel test — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 2.668, 95% CI 2-sided [0.923 to 7.710] — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: Phase 2: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), and Stable Disease (SD)
Description: DCR is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Up To 38 Months)
Population: Phase 2: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 81 | 86 | 46 | 43
Percentage of participants | 74.1 [63.1 to 83.2] | 72.1 [61.4 to 81.2] | 67.4 [52.0 to 80.5] | 62.8 [46.7 to 77.0]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Test type: Superiority; p = 0.7724, Exact Mantel-Haenszel test — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 1.106, 95% CI 2-sided [0.558 to 2.194] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Test type: Superiority; p = 0.6508, Exact Mantel-Haenszel test — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 1.222, 95% CI 2-sided [0.513 to 2.911] — [estimate comment as in outcome 2, analysis 1]

16. Secondary Outcome: Phase 2: Time to First Worsening of the Brief Pain Inventory Short Form Modified (mBPI-sf) "Worst Pain Score"
Description: The mBPI-sf is a 11-item instrument used as a multiple-item measure of cancer pain intensity ranging from 0 (no pain or does not interfere) and ranged through 10 (pain as bad as you can imagine or completely interferes). Time to first worsening of the mBPI-sf "worst pain score" (TWP) was defined as the time from the date of randomization to the first date of either a "worst pain" score increase of greater than or equal to (≥) 2 points from baseline or an analgesic drug class increase of ≥1 level. If the patient has not worsened by either of these criteria, TWP was censored for analysis on the last date the mBPI-sf was administered.
Time Frame: Baseline to Follow-up (Up To 24 Months)
Population: Phase 2: All randomized participants who had baseline and at least one post-baseline assessment (including the censored participants). Number of participants censored in "Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) = 30," "Placebo + Gemcitabine + Docetaxel (Olaratumab-naive)=23," "Olaratumab + Gemcitabine + Docetaxel (Olaratumab pre-treated)=17," "Placebo + Gemcitabine + Docetaxel (Olaratumab pre-treated)=8."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 68 | 71 | 41 | 34
Months | 3.61 [2.66 to 8.57] | 2.27 [1.41 to 6.54] | 3.15 [1.41 to 7.62] | 2.20 [0.76 to 3.02]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Test type: Superiority; p = 0.073, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.661, 95% CI 2-sided [0.419 to 1.041] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Test type: Superiority; p = 0.225, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.703, 95% CI 2-sided [0.395 to 1.253] — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: Phase 2: Time to First Worsening of Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) - Symptom Scales.
Description: The EORTC QLQ-C30 is a self-reported general cancer instrument consisting of 30 items covered by 1 of 3 dimensions: global health status/quality of life (2 items), functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, or financial impact). Time to first worsening of Symptom Burden was defined as the time from randomization to the first observation of worsening on symptom scales (i.e.,) increase of at least 10 points from baseline. For symptom scales, a linear transformation was used to obtain total score ranging from 0 to 100, a high score represents a high level of symptomatology or problems.
Time Frame: Baseline to Follow-up (Up to 33 months)
Population: Phase 2: All randomized participants who had baseline and at least one post-baseline assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 75 | 80 | 45 | 41
Months
  Fatigue: number analyzed (Participants) | 75 | 77 | 44 | 39
  Fatigue | 0.95 [0.76 to 1.12] | 0.95 [0.76 to 1.45] | 0.85 [0.72 to 1.41] | 0.76 [0.72 to 1.84]
  Nausea and vomiting: number analyzed (Participants) | 74 | 78 | 44 | 41
  Nausea and vomiting | 3.78 [2.14 to NA] — There were not enough events to estimate the upper confidence limit. | 2.46 [0.99 to 13.34] | 3.98 [1.41 to NA] — There were not enough events to estimate the upper confidence limit. | 13.17 [1.64 to NA] — There were not enough events to estimate the upper confidence limit.
  Pain: number analyzed (Participants) | 73 | 77 | 44 | 35
  Pain | 4.67 [2.33 to 9.53] | 0.99 [0.79 to 2.76] | 2.43 [1.41 to 8.77] | 3.06 [0.76 to 5.55]
  Dyspnoea: number analyzed (Participants) | 74 | 78 | 43 | 39
  Dyspnoea | 2.14 [1.51 to 3.06] | 2.14 [1.48 to 2.86] | 2.33 [1.45 to 14.09] | 2.79 [1.45 to 8.05]
  Insomnia: number analyzed (Participants) | 68 | 74 | 41 | 38
  Insomnia | 5.32 [2.33 to 7.72] | 4.24 [1.48 to 16.82] | 1.91 [1.41 to 6.47] | 5.09 [1.45 to NA] — There were not enough events to estimate the upper confidence limit.
  Appetite loss: number analyzed (Participants) | 73 | 76 | 45 | 37
  Appetite loss | 1.12 [0.82 to 2.14] | 2.56 [1.64 to 3.98] | 1.41 [0.85 to 3.52] | 1.97 [1.38 to 4.04]
  Constipation: number analyzed (Participants) | 73 | 77 | 44 | 40
  Constipation | 3.25 [2.14 to 5.98] | 2.86 [1.48 to NA] — There were not enough events to estimate the upper confidence limit. | 4.63 [1.91 to 12.91] | 3.81 [1.97 to NA] — There were not enough events to estimate the upper confidence limit.
  Diarrhoea: number analyzed (Participants) | 75 | 80 | 44 | 41
  Diarrhoea | 1.41 [0.99 to 3.68] | 1.81 [1.41 to 4.24] | 3.55 [1.41 to 6.05] | 3.52 [1.97 to NA] — There were not enough events to estimate the upper confidence limit.
  Financial difficulties: number analyzed (Participants) | 67 | 71 | 43 | 35
  Financial difficulties | NA [5.32 to NA] — There were not enough events to estimate the median, upper confidence limit. | 7.66 [3.29 to NA] — There were not enough events to estimate the upper confidence limit. | 7.29 [2.33 to 7.85] | NA [3.94 to NA] — There were not enough events to estimate the upper confidence limit.
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Fatigue; Test type: Superiority; p = 0.332, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.213, 95% CI 2-sided [0.834 to 1.764] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Nausea and vomiting; Test type: Superiority; p = 0.389, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.813, 95% CI 2-sided [0.514 to 1.287] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Pain; Test type: Superiority; p = 0.020, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.598, 95% CI 2-sided [0.386 to 0.926] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Dyspnoea; Test type: Superiority; p = 0.821, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.947, 95% CI 2-sided [0.622 to 1.442] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Insomnia; Test type: Superiority; p = 0.812, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.931, 95% CI 2-sided [0.574 to 1.509] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Appetite loss; Test type: Superiority; p = 0.162, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.355, 95% CI 2-sided [0.893 to 2.055] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Constipation; Test type: Superiority; p = 0.619, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.881, 95% CI 2-sided [0.550 to 1.413] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Diarrhoea; Test type: Superiority; p = 0.597, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.134, 95% CI 2-sided [0.746 to 1.724] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive); Financial difficulties; Test type: Superiority; p = 0.380, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.766, 95% CI 2-sided [0.425 to 1.381] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Fatigue; Test type: Superiority; p = 0.877, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.046, 95% CI 2-sided [0.635 to 1.723] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Nausea and vomiting; Test type: Superiority; p = 0.791, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.102, 95% CI 2-sided [0.568 to 2.139] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Pain; Test type: Superiority; p = 0.487, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 0.810, 95% CI 2-sided [0.454 to 1.443] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Dyspnoea; Test type: Superiority; p = 0.976, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.014, 95% CI 2-sided [0.556 to 1.850] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Insomnia; Test type: Superiority; p = 0.111, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.694, 95% CI 2-sided [0.882 to 3.250] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Appetite loss; Test type: Superiority; p = 0.760, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.108, 95% CI 2-sided [0.620 to 1.979] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Constipation; Test type: Superiority; p = 0.747, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.119, 95% CI 2-sided [0.586 to 2.135] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Diarrhoea; Test type: Superiority; p = 0.330, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.367, 95% CI 2-sided [0.726 to 2.576] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) vs Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated); Financial difficulties; Test type: Superiority; p = 0.411, Log Rank — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.373, 95% CI 2-sided [0.636 to 2.965] — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: Phase 2: Health Status on the EuroQol 5-Dimension 5 Level (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) of health status are each assessed with 5 response options (1=no problem, 2=slight, 3=moderate, 4=severe, and 5=extreme problem) and scored as a composite index which were anchored on a scale of 0 to 1 with a higher score representing better health status. Additionally, current health status was assessed on a visual analogue scale (VAS) ranging from 0 to 100 with a higher score representing better health status.
Time Frame: Cycle 1 (Day 1), Follow-up (Up to 38 Months)
Population: Phase 2: All randomized participants who completed EQ-5D-5L.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 71 | 75 | 42 | 35
score on a scale
  EQ-5D-5L - Index Value [Cycle 1 (Day 1)]: number analyzed (Participants) | 71 | 74 | 39 | 35
  EQ-5D-5L - Index Value [Cycle 1 (Day 1)] | 0.80 (0.17) | 0.81 (0.17) | 0.83 (0.15) | 0.83 (0.22)
  EQ-5D-5L - VAS Score [Cycle 1 (Day 1)] | 73.5 (18.9) | 72.7 (18.1) | 76.2 (19.6) | 70.3 (23.8)
  EQ-5D-5L - Index Value [Follow-up (Up to 38 Months)]: number analyzed (Participants) | 42 | 50 | 26 | 25
  EQ-5D-5L - Index Value [Follow-up (Up to 38 Months)] | 0.74 (0.21) | 0.71 (0.26) | 0.80 (0.20) | 0.76 (0.24)
  EQ-5D-5L - VAS Score [Follow-up (Up to 38 Months)]: number analyzed (Participants) | 42 | 50 | 26 | 25
  EQ-5D-5L - VAS Score [Follow-up (Up to 38 Months)] | 68.7 (16.5) | 63.0 (21.6) | 74.8 (21.8) | 70.8 (24.2)

19. Secondary Outcome: Phase 2: Number of Participants With Treatment Emergent Anti-Olaratumab Antibodies
Description: Number of Participants with Treatment Emergent Anti-Olaratumab Antibodies
Time Frame: Baseline through Follow-Up (Up to 38 Months)
Population: Phase 2: All randomized participants who received at least one dose of Olaratumab and had evaluable immunogenicity data.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
Number analyzed (Participants) | 77 | 43
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 38 Months)
Description: Phase 1b/2: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated)
All-Cause Mortality (participants affected / at risk) | 15/21 | 11/18 | 12/15 | 54/81 | 28/45 | 58/86 | 28/43
Serious Adverse Events (participants affected / at risk) | 6/21 | 9/18 | 9/15 | 44/81 | 21/45 | 38/86 | 23/43
Other Adverse Events (participants affected / at risk) | 21/21 | 18/18 | 15/15 | 78/81 | 45/45 | 81/86 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel (N=21) | Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel (N=18) | Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel (N=15) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) (N=81) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) (N=45) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) (N=86) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated) (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 2 (2) | 4 (5) | 0 (0)
Bandaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 3 (3) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (5) | 3 (5) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 2 (2) | 7 (8) | 6 (6)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 6 (6) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1b: Cohort 1 - 15 mg/kg Olaratumab + Gemcitabine + Docetaxel (N=21) | Phase 1b: Cohort 2 - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel (N=18) | Phase 1b: Cohort 2 Expansion - 20 mg/kg Olaratumab + Gemcitabine + Docetaxel (N=15) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab-naive) (N=81) | Phase 2: Olaratumab + Gemcitabine + Docetaxel (Olaratumab Pre-treated) (N=45) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab-naive) (N=86) | Phase 2: Placebo + Gemcitabine + Docetaxel (Olaratumab Pre-treated) (N=43)
Anaemia (Blood and lymphatic system disorders) | 13 (42) | 12 (54) | 9 (24) | 43 (168) | 33 (145) | 47 (147) | 20 (57)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (13) | 1 (4) | 3 (6) | 1 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 3 (4) | 2 (5) | 20 (55) | 6 (6) | 24 (43) | 4 (10)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (8) | 3 (3) | 4 (12) | 10 (21) | 9 (18) | 13 (21) | 6 (12)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 3 (3) | 5 (8) | 2 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 3 (3) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 3 (3) | 3 (3)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 9 (11) | 7 (12) | 10 (10) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 2 (2) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (8) | 3 (7) | 4 (6) | 21 (29) | 12 (14) | 20 (24) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 7 (22) | 8 (14) | 5 (8) | 36 (84) | 21 (42) | 30 (50) | 14 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (6) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2) | 6 (9) | 2 (2) | 8 (9) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 6 (7) | 5 (5) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 9 (15) | 3 (4) | 38 (59) | 20 (31) | 40 (73) | 12 (22)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (8) | 1 (1) | 0 (0) | 17 (34) | 7 (18) | 15 (26) | 11 (20)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2) | 1 (1) | 25 (30) | 7 (8) | 13 (17) | 7 (13)
Asthenia (General disorders) | 4 (21) | 2 (8) | 0 (0) | 12 (59) | 1 (1) | 14 (58) | 3 (9)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (3) | 1 (1) | 8 (13) | 5 (5) | 4 (5) | 7 (8)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (32) | 14 (35) | 12 (21) | 49 (126) | 34 (76) | 45 (110) | 23 (44)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 3 (6) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 7 (9) | 3 (4) | 8 (8) | 3 (3)
Non-pitting oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 8 (13) | 5 (9) | 5 (8) | 37 (67) | 21 (36) | 23 (33) | 14 (21)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (2) | 8 (11) | 0 (0)
Pyrexia (General disorders) | 6 (8) | 8 (11) | 2 (2) | 23 (51) | 10 (12) | 26 (49) | 11 (17)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 3 (4) | 3 (4)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 5 (6) | 2 (2) | 3 (4)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 1 (1) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 7 (9) | 3 (4) | 14 (19) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 15 (18) | 3 (4) | 8 (8) | 1 (1)
Vaginal infection (Infections and infestations) | 0/11 (0) | 0/8 (0) | 1/7 (1) | 0/48 (0) | 0/28 (0) | 0/58 (0) | 0/28 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 2 (3) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (7) | 6 (13) | 2 (2) | 13 (36) | 8 (19) | 16 (33) | 7 (20)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 4 (7) | 2 (2) | 10 (22) | 6 (15) | 11 (14) | 3 (7)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 3 (6) | 2 (2) | 7 (15) | 11 (22) | 4 (6) | 3 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (6) | 3 (3) | 4 (4) | 2 (9)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (5) | 3 (5) | 0 (0) | 4 (5) | 4 (4) | 1 (4) | 3 (5)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 4 (15) | 0 (0) | 8 (31) | 5 (32) | 9 (33) | 3 (4)
Neutrophil count decreased (Investigations) | 1 (3) | 5 (7) | 0 (0) | 16 (44) | 20 (72) | 14 (32) | 4 (4)
Platelet count decreased (Investigations) | 2 (2) | 7 (15) | 2 (2) | 19 (50) | 15 (44) | 16 (46) | 7 (10)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 4 (6) | 0 (0) | 5 (9) | 3 (4) | 6 (14) | 5 (7)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 7 (11) | 0 (0) | 1 (1) | 1 (2)
White blood cell count decreased (Investigations) | 3 (3) | 4 (11) | 0 (0) | 12 (50) | 12 (63) | 12 (43) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 6 (8) | 0 (0) | 21 (33) | 11 (14) | 15 (30) | 14 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 3 (4) | 2 (2) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (5) | 0 (0) | 6 (7) | 10 (16) | 4 (4) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0) | 8 (9) | 4 (6) | 2 (3) | 5 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 5 (6) | 4 (5) | 1 (1) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (10) | 1 (1) | 6 (10) | 9 (16) | 10 (24) | 7 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 3 (5) | 3 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (8) | 3 (4) | 0 (0) | 4 (7) | 2 (2) | 2 (7) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (6) | 1 (1) | 4 (8) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 2 (3) | 13 (24) | 6 (8) | 14 (18) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (7) | 6 (7) | 10 (16) | 7 (8) | 7 (10) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 9 (10) | 5 (5) | 7 (7) | 6 (6)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 3 (4) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 6 (9) | 7 (8) | 5 (10) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (6) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 6 (6) | 4 (4) | 16 (27) | 13 (16) | 11 (18) | 11 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 1 (1) | 13 (16) | 5 (7) | 8 (9) | 4 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (4) | 11 (26) | 3 (4) | 9 (12) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (7) | 7 (7) | 0 (0) | 12 (20) | 13 (21) | 11 (11) | 14 (18)
Headache (Nervous system disorders) | 5 (6) | 5 (5) | 1 (1) | 15 (23) | 6 (7) | 13 (15) | 5 (5)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 7 (10) | 0 (0) | 5 (5) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 4 (4) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (6) | 1 (2) | 3 (8) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 10 (15) | 10 (20) | 13 (31) | 9 (14)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (6) | 3 (3)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (5) | 2 (2) | 5 (5) | 2 (2) | 5 (5) | 3 (4)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 15 (17) | 6 (7) | 7 (8) | 10 (11)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 1 (3) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (9) | 1 (3) | 16 (22) | 13 (21) | 21 (27) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (11) | 5 (9) | 19 (30) | 15 (30) | 18 (25) | 12 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 5 (7) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (5) | 16 (19) | 5 (6) | 17 (22) | 9 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (3)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 4 (4) | 6 (6) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (4) | 6 (7) | 1 (1) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 3 (3) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 5 (6) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (10) | 1 (1) | 29 (35) | 5 (5) | 32 (44) | 5 (5)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 4 (5) | 2 (3) | 2 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 5 (5) | 5 (6) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 5 (6) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 3 (3) | 4 (4) | 2 (3)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 3 (3) | 2 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 6 (16) | 3 (8) | 4 (7) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 2 (3) | 6 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 15 (17) | 1 (1) | 11 (17) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 10 (17) | 6 (7) | 6 (7) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (3) | 4 (4) | 0 (0)
Orchidectomy (Surgical and medical procedures) | 0/10 (0) | 0/10 (0) | 1/8 (1) | 0/33 (0) | 0/17 (0) | 0/28 (0) | 0/15 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 2 (2)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 10 (13) | 2 (2) | 4 (7) | 5 (6)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 5 (9) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (20) | 6 (6) | 7 (23) | 6 (7)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 8 (8) | 5 (5) | 2 (2)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02659020/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT02659020/SAP_001.pdf